CLINICAL TRIAL: NCT02301767
Title: MRI Background Parenchymal Enhancement as a Risk Factor for Breast Cancer: The IMAGINg and Epidemiology (IMAGINE) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Pennsylvania (Other); University of Utah (Other); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-246
Record Dates: First submitted 2014-11-19; First posted 2014-11-26 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: MRI; Risk Factor; background Parenchymal Enhancement; (IMAGINE) Study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva

GROUPS / COHORTS (2):
- women that are diagnosed with breast cancer: To complete the study women need to have undergone their scheduled contrast-enhanced MRI, completed the study questionnaire, and provided written consent to release MRIs/mammograms. Although attempts will be made to obtain written consent from all women, the questionnaire data captured from the women who only provide verbal consent may be used in analysis. Optional saliva samples will also be collected for future use.
- women at high risk of breast cancer: To complete the study women need to have undergone their scheduled contrast-enhanced MRI, completed the study questionnaire, and provided written consent to release MRIs/mammograms. Although attempts will be made to obtain written consent from all women, the questionnaire data captured from the women who only provide verbal consent may be used in analysis. Optional saliva samples will also be collected for future use.

SUMMARY:
The purpose of the study is to view what normal breast tissue looks like on an MRI and mammogram to help determine how it may affect the risk of developing breast cancer. The investigators will also compare the information collected from the questionnaire and medical records to help better understand how this may affect the risk of developing breast cancer. If a saliva or tissue sample is collected for future use, this information will enable us to study genetic risk factors as well.

DETAILED DESCRIPTION:
Proposed Study Methods Pertaining to the Population, Eligibility and Recruitment In this multi-center hospital-based case-control study, cases will be women diagnosed with incident breast cancer who have undergone or are about to undergo a bilateral breast MRI with contrast to assess extent of disease. The cancer-free controls will be women at high-risk of breast cancer undergoing a bilateral breast MRI with contrast for screening. The MRI collected for the study may be post-biopsy and post-surgery (unilateral lumpectomy/mastectomy), but prior to bilateral mastectomy, radiation, hormonal, and/or chemotherapy. Study participants also need to have a bilateral mammogram available at the study site within 24 months prior to, or up to 24 months after the study MRI (as long as prior to surgery, radiation, hormonal, and/or chemotherapy), to be included in the secondary aim analysis. The MRI/mammogram selected for this study do not need to be conducted at the recruitment site, the digital images just need to be accessible from the patient medical records at the site. Questionnaire data, optional saliva samples, MRIs, mammograms, and medical records will be collected over a 27 month period from women at three NCI-designated comprehensive cancer centers (MSK, Penn, Utah). Each site has demonstrated experience with recruitment, patient interviews and collection of MRIs and mammograms.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria for Breast Cancer Cases (invasive)

Women with the following characteristics at MRI will be eligible as invasive cases:

1. have a diagnosed invasive unilateral breast cancer after 1/1/2010;
2. have a pre-treatment (prior to bilateral mastectomy, radiation, hormonal, and/or chemotherapy) bilateral breast MRI with contrast available from the study site;
3. be ≥ 21 and <70 years old at time of diagnosis; and
4. have an intact contralateral breast at the time of study MRI.

Eligibility Criteria for Breast Cancer Cases (non-invasive)

Women with the following characteristics at MRI will be eligible as non-invasive cases:

have a diagnosed unilateral ductal carcinoma in situ (DCIS) preferably after 1/1/2013; 2) have a pre-treatment (prior to bilateral mastectomy, radiation, hormonal, and/or chemotherapy) bilateral breast MRI with contrast available from the study site; 3) be ≥ 21 and <70 years old at time of diagnosis; and 4) have an intact contralateral breast. The contralateral breast needs to be intact and unaffected by an invasive carcinoma and/or DCIS so the MRI reading can be done on the breast without cancer. Women with a history of previous cancer diagnosis are excluded because treatment they may have received for these cancers might affect the MRI readings.

Eligibility Criteria for Controls Controls will be women determined to be at high risk of developing breast cancer (i.e., lifetime risk ≥20%

Controls must meet the following criteria:

1. have a bilateral breast MRI screening with contrast available from the study site;
2. be ≥ 21 and <70 years old at time of MRI; and
3. negative breast MRI screen.

Exclusion Criteria:

* For either cases or controls prior to study MRI date:

  1. unable to speak and read English;
  2. history of prophylactic mastectomy;
  3. history of pre-pectoral breast implants in either breast (sub-pectoral are acceptable);
  4. history of breast reduction surgery;
  5. currently taking, or in the previous 3 months: hormonal medication such as Tamoxifen (Nolvadex), Raloxifene (Evista), aromatase inhibitors (Anastrozole/Arimidex, Letrozole/Femara, and/or Exemestane/Aromasin); and/or other postmenopausal hormonal therapy (PHT) medication; and/or hormonal medication for fertility treatment; [Note: Women are INELIGIBLE if they report taking pills orally, use a patch or ring, even if just intermittently used. Women are ELIGIBLE if they report just taking hormone replacement therapy in the form of a cream, suppository (or intra-vaginal), soy-based, or other natural product.]
  6. currently, or in the preceding 6 months, pregnant or breast feeding; and
  7. history of previous cancer including DCIS [Note: Women are ELIGIBLE if diagnosed with non melanoma skin cancer lobular carcinoma in situ (LCIS) and/or cervical cancer in situ ].

Notes: Women recently diagnosed with DCIS within the study period will be categorized as non-invasive cases (preferable prospective recruitment only). Only one breast may be affected by a recent diagnosis of invasive carcinoma and/or DCIS.

Ages: 21 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The three data cancer centers (MSK, Penn, Utah) will recruit 1,110 cases (women diagnosed with breast cancer) and 1,110 matched controls (high risk women).
Sampling Method: Non-Probability Sample
Enrollment: 2187 (Actual)
Dates: Start 2014-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Case/control status | 2 years

SECONDARY OUTCOMES:
Complete questionnaires | 2 years
MRI-BPE measurements | 2 years
MRI-FGT measurements | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonine Bernstein, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Watt GP, Thakran S, Sung JS, Jochelson MS, Lobbes MBI, Weinstein SP, Bradbury AR, Buys SS, Morris EA, Apte A, Patel P, Woods M, Liang X, Pike MC, Kontos D, Bernstein JL. Association of Breast Cancer Odds with Background Parenchymal Enhancement Quantified Using a Fully Automated Method at MRI: The IMAGINE Study. Radiology. 2023 Sep;308(3):e230367. doi: 10.1148/radiol.230367. PMID 37750771
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02301767/ICF_000.pdf